CLINICAL TRIAL: NCT01091181
Title: The Effect of Hysterotomy Technique on the Rate of Large Defects in the Hysterotomy Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2-valentin; NCT03498339 (obsolete NCT alias)
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Scars
Keywords: Caesarean
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: women aimed for emergency cesarean section were randomized into two groups according to surgery technique of opening the uterus: 1 Group - high level of hysterotomy incision; 2 Group - low level of hysterotomy incision. Opening and closing of abdomen performed in the same manner in both groups
Who Masked: Participant, Investigator
Masking Description: the surgeon who performed the operation knew what technique to use. Participant were not informed in what group they were. Six months postpartum patients came to ultrasound department and underwent ultrasound examination of uterus and uterine cesarean scar. Sonographer was blinded to the surgery technique.
Oversight: Data Monitoring Committee: No

ARMS (2):
- high incision group (Active Comparator): hysterotomy at cesarean performed 2 cm above plica vesicouterina
  Interventions: Procedure: hysterotomy at cesarean
- low incision group (Active Comparator): hysterotomy at cesarean performed 2 cm below plica vesicouterina
  Interventions: Procedure: hysterotomy at cesarean

INTERVENTIONS:
Procedure: hysterotomy at cesarean — incision to open the uterus at cesarean.

SUMMARY:
The Effect of Cesarean Operative Technique on the Occurrence of Large Hysterotomy Scar Defects.

DETAILED DESCRIPTION:
Having a Caesarean leads to a scar in the uterus, which does not always heal properly. Defective healing can lead to serious complications in the next pregnancy and delivery. Different surgical techniques can be used for a Caesarean section.

The aim is to compare two surgical techniques (different ways of opening the uterus), to investigate whether one or the other technique leads to fewer defective scars in the uterus. Both these techniques are in use at the clinic. After the operation, patients are cared for in the normal way.

Six months after the Caesarean, patients are examined using vaginal ultrasound. Vaginal ultrasound allows to see if the scar after the Caesarean has healed well, or if there are defects in it.

ELIGIBILITY:
inclusion criteria:

* ≥ 18 years old
* gestational age ≥ 37 gestational weeks
* cervical dilatation ≥5 cm,
* no previous uterine surgery other than cone biopsy, loop electrosurgical excision procedure, dilatation and curettage, or dilatation and evacuation, undergoing emergency caesarean section.

exclusion criteria:

• need of immediate caesarean section, defined as delivery of the baby within 20 minutes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
large defect | 6 months
  occurrence of large defects in uterine cesarean scar are detected by ultrasound and are assessed by the percentage of patients who have large defects in uterine cesarean scar

SECONDARY OUTCOMES:
APGAR score | 1 and 5 minute after delivery
  APGAR score measured at 1 and 5 minute after delivery. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10.
blood loss | 1 hour
  estimated blood loss during surgery is measured in terms of mL
difficulties at delivery of fetus | 1 hour
  difficulties at delivery of fetus at caesarean are assessed by the percentage of patients when surgeons experience difficulties at delivery of fetus at caesarean
postoperative infection | 8 weeks
  postoperative infection after caesarean section is assessed by the percentage of patients who develop this complication
readmission to the hospital | 8 weeks
  readmission to the hospital due to need of re-operation is assessed by the percentage of patients who have re-operation after caesarean
miscarriage | up to 8 years
  occurrence of miscarriage in subsequent pregnancy is assessed by the percentage of patients who have miscarriages in subsequent pregnancy
scar pregnancy | up to 8 years
  occurrence of scar pregnancy in subsequent pregnancy is assessed by the percentage of patients who have scar pregnancy after the index caesarean
placenta previa/accreta | up to 8 years
  occurrence of placenta previa/accreta in subsequent pregnancy is assessed by the percentage of patients who have placenta previa/accreta in subsequent pregnancy
uterina rupture/uterine dehiscence | up to 8 years
  occurrence of uterine rupture/uterine dehiscence in subsequent labour is assessed by the percentage of patients who have uterine rupture/uterine dehiscence in subsequent labour
vaginal delivery after caesarean | up to 8 years
  success rate of vaginal delivery after caesarean is assessed by the percentage of patients who delivered vaginally after the index caesarean

CONTACTS AND LOCATIONS:
Overall Officials: Olga Vikhareva, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skåne University Hospital Malmö, Malmo, Sweden